CLINICAL TRIAL: NCT01590693
Title: Botulinum Toxin A Does Not Improve Cast Treatment for Idiopathic Toe-walking- a Prospective Randomized Trial.
Brief Title: Botulinum Toxin A for Idiopathic Toe-walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pahr Engstrom, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S4
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Idiopathic Toe-walking
Keywords: Gait
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Experimental): Children treated with four weeks of below knee walking casts and botulinum toxin A injections
  Interventions: Drug: Botulinum toxin A
- Group 1 (Active Comparator): Children treated with four weeks of below knee walking casts.
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — The children in Group 2 underwent bilateral treatment with a total of 12 units/kg bodyweight Botox® (Allergan, California, USA). Four injection sites in each calf - two in the proximal third of the lateral and medial gastrocnemius bellies and two distally in the gastrocnemius-soleus complex - were administered. All injections were performed with electromyogram amplifier guidance to ensure intramuscular position. Children in both groups were treated with four weeks of below knee walking casts. Children in group 2 received the casts 1-2 weeks after botulinum toxin A treatment.

SUMMARY:
The purpose of this study is to determine whether botulinum toxin A (BTX) adds a favourable effect to treatment of idiopathic toe-walking with below knee walking casts. The specific hypothesis to be tested is that a combination of BTX and casting is more effective than casting treatment alone in reducing toe-walking in 5-15 year old children. Evaluation methods include 3-D gait analysis, parents' perception of toe-walking frequency, passive joint range of motion measurements, and strength of ankle dorsal extension.

ELIGIBILITY:
Inclusion Criteria:

* Children with idiopathic toe-walking
* 5-15 years of age

Exclusion Criteria:

* Previous treatment for idiopathic toe-walking, such as, Achilles tendon surgery, casting, orthotics, and BTX treatment.
* Flexion contracture beyond -10 degrees in the ankle

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2005-11; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of toe-walking | baseline, 3month, 12 month

SECONDARY OUTCOMES:
Joint range of movement | Baseline, 3 month, 12 month
Classification of idiopathic toe-walking | Baseline, 3 month, 12 month
Gait analysis parameters | Baseline, 3 month, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Pähr Engstrom, MD., Dr., Principal Investigator — Karolinska Institutet
Locations (1):
- Astrid Lindren Children's Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Engstrom P, Bartonek A, Tedroff K, Orefelt C, Haglund-Akerlind Y, Gutierrez-Farewik EM. Botulinum toxin A does not improve the results of cast treatment for idiopathic toe-walking: a randomized controlled trial. J Bone Joint Surg Am. 2013 Mar 6;95(5):400-7. doi: 10.2106/JBJS.L.00889. PMID 23467862